CLINICAL TRIAL: NCT06635200
Title: Determination of Dominant Pain Phenotype in Patients With Carpal Tunnel Syndrome
Brief Title: Pain Phenotype in Patients With Carpal Tunnel Syndrome
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Emrah Afsar, Phd, Kutahya Health Sciences University
Other Study IDs: 2024
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with carpal tunnel syndrome with a nociceptive pain phenotype
- Patients with carpal tunnel syndrome with a neuropathic pain phenotype
- Patients with carpal tunnel syndrome with a nosiplastic pain phenotype

SUMMARY:
The aim of this study was to determine the dominant pain phenotype in a group of patients with Carpal Tunnel Syndrome by applying the International Association for the Study of Pain (IASP) criteria.

DETAILED DESCRIPTION:
Voluntary participants between the ages of 18-65 who have been diagnosed with CTS will be included in the study.The 7 steps in the Clinical Criteria/Rating System determined by the International Association for the Study of Pain (IASP) for Nosiplastic Pain and Carpal Tunnel Syndrome will be applied to people with CTS. Thermal pain threshold, mechanical pain sensitivity and static/dynamic allodynia will be evaluated to determine pain hypersensitivity (Step 5). Specific questions will be asked to confirm the history of hypersensitivity in patients (Step 6). Finally, comorbidities, if any, will be determined (Step 7). As a result, the pain phenotype of patients with CTS will be determined (Nociceptive, Neuropathic or Nosiplastic). Shapiro-Wilk test will be performed to determine the distribution of the data. One-way ANOVA (continuous) or Kruskal-Wallis (categorical) will be used to examine whether the dependent variables differ between groups. For significant F-test, an additional investigation of differences between groups will be performed with Gabriel's post hoc procedure.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with CTS
* Being between the ages of 18-65
* Volunteering to participate in the study

Exclusion Criteria:

* Having systemic inflammatory disease
* Having a disease that may cause polyneuropathy such as diabetes mellitus
* Having a pacemaker
* Having a disease affecting the central nervous system
* Having cervical radiculopathy
* History of previous operation or local steroid injection due to CTS
* Hypersensitivity to heat and cold

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Voluntary participants between the ages of 18-65 who have been diagnosed with Carpal Tunnel Syndrome will be included in the study
Sampling Method: Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-03-18 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale | 1 minute
  Patients rate the current pain intensity from 0 ("no pain") to 10 ("worst possible pain").

SECONDARY OUTCOMES:
Cold Pain Threshold | 2 minutes
  For cold pain threshold, ice cubes (-5°C) placed in a plastic bag will be placed on the patients' skin for 10 seconds. Increased sensory perception will be considered as gain of function. The intensity of pain will also be recorded on an NRS scale ranging from 0 (no pain) to 10 (worst pain imaginable).
Hot Pain Threshold | 2 minutes
  Thermal pain perception will be tested using a 3 cm2 sized metal piece equal to (lab-QST thermode size). The metal parts will be heated to 45˚C for hot pain threshold. The metal pieces will be applied to the skin for 3 seconds. It will be determined whether the stimulus is painful (yes/no), and if painful, the intensity of the pain on a numerical rating scale (NRS) (0: no pain, 10: imaginably worse pain).
Mechanical Pain Threshold | 3 minutes
  Mechanical pain threshold: to be assessed with a toothpick and a von Frey filament (256 mN). Increased sensory perception will be considered to reflect gain of function. The intensity of pain will also be recorded on an NRS scale ranging from 0 (no pain at all) to 10 (worst pain imaginable).
Static mechanical allodynia | 3 minutes
  A digital algometer will be used to measure Pressure Pain Threshold levels. Pressure will be applied at a rate of approximately 30 kPa with the algometer placed perpendicular to the point of application. Participants will be instructed to report when the sensation changes from pressure to pain. The intensity of pain will also be recorded on an NRS scale ranging from 0 (no pain at all) to 10 (worst pain imaginable).
Dynamic Mechanical Allodynia | 3 minutes
  Patients will be touched on the affected area and the control area with a brush, an ear stick and a piece of cotton wool. The assessment tools will be applied 4 times by drawing a cross of 2 strokes (length 5 cm) at an angle of 90˚C in each direction. For each stimulus (brush/ear swab/cotton swab), they will indicate (1) whether the stimulus was perceived as painful (yes/no) and (2) the pain intensity on the NRS-11 (0 no pain, 10 imaginably worse pain).

CONTACTS AND LOCATIONS:
Overall Officials: Emrah Afsar, Phd, Principal Investigator — Kutahya Health Science University
Locations (1):
- Kutahya Health Science University, Kütahya, Turkey (Türkiye)